CLINICAL TRIAL: NCT03971656
Title: Preoperative Nutritional Intervention in Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00143484
Record Dates: First submitted 2019-05-24; First posted 2019-06-03 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Head and Neck Cancer; Malnutrition
Keywords: Cancer; Surgery; Malnutrition; Preoperative; Nutrition
MeSH Terms: conditions — Head and Neck Neoplasms; Malnutrition; Neoplasms | interventions — Dietary Supplements; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard care
- Intervention (Experimental): Three-Fold Nutritional Intervention
  Interventions: Dietary Supplement: Nutritional Supplement; Behavioral: Preoperative Dietitian Consult; Behavioral: Education

INTERVENTIONS:
Dietary Supplement: Nutritional Supplement — Oral nutritional supplementation
  Arms: Intervention
Behavioral: Preoperative Dietitian Consult — Nutritional assessment
  Arms: Intervention
Behavioral: Education — Informational materials about nutrition
  Arms: Intervention

SUMMARY:
The purpose of this study is to determine the impact of preoperative nutritional supplements on head and neck surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 who are seen in the Department of Otolaryngology-Head and Neck Surgery clinic, have a new H&N cancer diagnosis, and have not undergone previous treatment for H&N cancer are eligible for this study. We will enroll only patients who will be undergoing primary surgery for their cancer treatment, and those undergoing primary radiation or primary chemoradiation for treatment will be excluded. All eligible patients will undergo nutritional screening using the PG-SGA. Those who screen positive for malnutrition (>1 on the PG-SGA scale) will be randomized to either our standard care (control) versus nutritional intervention group.

Exclusion Criteria:

* Prior treatment for head and neck cancer. Those undergoing primary radiation or chemoradiation for their head and neck cancer. Vulnerable populations. Patients who screen as well nourished (>1 on the PG-SGA scale) will be excluded as they do not require nutritional intervention. Patients who screen as severely malnourished (>8 on the PG-SGA scale) will be excluded as these patients require intervention and should not be potentially randomized to our control arm. Patients requiring nasogastric tube feeding or gastrostomy tube feeding will be excluded. Patients are routinely evaluated by speech pathologist prior to surgery. Those in which there is concern for aspiration will be excluded as they will not be able to participate fully in the intervention.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2020-12-11 (Actual); Study Completion 2022-10-17 (Actual)

PRIMARY OUTCOMES:
Change in Scored Patient-Generated Subjective Global Assessment | Baseline and day of surgery
  PG-SGA is an interdisciplinary patient assessment of weight, intake, symptoms, functional status, disease state, metabolic stress and nutritional physical examination

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No